CLINICAL TRIAL: NCT02639572
Title: Evaluation of the Efficacy of a Novel Synthetic Bone Regeneration Material (Sil-Oss®) In the Treatment of Periodontal Intrabony Osseous Defects
Brief Title: Evaluation of SilOss® in Periodontal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SVS Institute of Dental Sciences (Other)
Collaborators: AzureBio, Madrid, Soain (Unknown)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Professor and Head, Periodontics, SVSIDS, Mahabubnagar, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/1/2014; Reg.no. D139406039 (Other: Dr NTR University of Health Sciences, Vijayawada, India)
Record Dates: First submitted 2015-12-20; First posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Siloss® bone graft (Experimental): Based on the sequence, in the test site,Siloss® was placed.
  Interventions: Biological: Siloss® bone graft
- Hydroxyapatitie Bone graf (Placebo Comparator): Based on the sequence, the control site which was treated by Hydroxyapatite graft only.
  Interventions: Biological: Hydroxyapatitie Bone graft

INTERVENTIONS:
Biological: Siloss® bone graft — The osseous defect was debrided of granulation tissue and the root surface was planed to remove plaque and calculus, until a smooth hard consistency was found. The defect's architecture was confirmed by direct observation and classified based on number of bony walls present. In patients selected for test group, in addition to open flap debridement (OFD), Siloss® bone replacement graft was utilized to fill the defects to the most coronal level of the osseous walls. The required amount of composite alloplast (Siloss®) was dispensed into a sterile dappen dish and mixed with patients own blood and carried to the defect site with an amalgam carrier. The mucoperiosteal flaps were repositioned and secured in place using interrupted sutures. The surgical procedure in control site included open flap debridement followed by placement of hydroxyapatite graft (G-graft®, Saharanpur, UP, India). The surgical area was protected and covered using a periodontal dressing. Randomization was employed.
  Arms: Siloss® bone graft
Biological: Hydroxyapatitie Bone graft — The osseous defect was debrided of granulation tissue and the root surface was planed to remove plaque and calculus, until a smooth hard consistency was found. The defect's architecture was confirmed by direct observation and classified based on number of bony walls present. In patients selected for test group, in addition to open flap debridement (OFD), Siloss® bone replacement graft was utilized to fill the defects to the most coronal level of the osseous walls. The required amount of composite alloplast (Siloss®) was dispensed into a sterile dappen dish and mixed with patients own blood and carried to the defect site with an amalgam carrier. The mucoperiosteal flaps were repositioned and secured in place using interrupted sutures. The surgical procedure in control site included open flap debridement followed by placement of hydroxyapatite graft (G-graft®, Saharanpur, UP, India). The surgical area was protected and covered using a periodontal dressing.Randomization was employed.
  Arms: Hydroxyapatitie Bone graf

SUMMARY:
Siloss® (Azurebio, Madrid, Spain) is a synthetic and inorganic bone graft material and is composed of a dicalcium phosphate anhydrous (monetite), hydroxyapatite (HA), and amorphous silica and trace amounts of zinc. It is manufactured by a proprietary process avoiding high temperatures. This results in a non-sintered material with a high specific surface area (65 m2/g) and high interconnected porosity (60%) that favour a high degree of interaction with its biological surrounding. It is fully resorbable, being replaced by natural bone, thereby avoiding the disadvantages of nonresorbable materials that interfere with normal processes of bone remodelling. Siloss® is resorbed both by a dual process of slow dissolution of its components and by active cellular remodelling. Controlled dissolution of Siloss® releases Ca, P, Si and Zn that stimulate regeneration processes while larger pores are formed allowing colonization of osteoclasts and osteoblasts involved in bone remodelling. It functions as a bioactive temporary scaffold maintaining the desired volume while it promotes bone regeneration and is being replaced by new vascularized bone. The alloplastic property of the graft material avoids the risk of infection and adverse inflammatory reactions. Also, resorption of Siloss® prevents possible adverse effects associated with long permanence of low resorbable materials.

The aim of the present study is to clinically and radiographically evaluate the efficacy of bone graft material (Siloss ®) in the treatment of intrabony defects.

DETAILED DESCRIPTION:
Study design The study was designed as a split-mouth, double-blind, randomized controlled clinical trial. The purpose of this study is to evaluate the efficacy of a novel synthetic bone regeneration material (Siloss®) in the treatment of periodontal intrabony osseous defects. Ethical clearance has been obtained from the institutional ethical committee with participants signing an informed consent prior to the commencement of the study.

Sample Size calculation Sample size was calculated by considering this trial as a non-inferiority trial. A minimum sample size of 27 will be required when the minimum difference of mean bone fill levels before and after treatment is to be at least 1mm2 at p=0.05 with expected variance of 0.8 for having ß=0.1.

Source of data A total of 30 subjects were selected from the outpatient section of the Department of Periodontics. Systemically healthy chronic periodontitis subjects within the age group of 30-55 years having at least 2 periodontal pockets ≥5 mm with at least 1 pocket in each quadrant showing ra¬diographic evidence of vertical bone loss were included in the study. Patients who underwent periodontal therapy in the past 6 months and/or have used antibiotic drugs, antioxidants, and antibacterial mouthwash or medicated toothpastes within 6 months of baseline and smokers were excluded from the study. Assessment of suitability for bone graft was confirmed by transgingival probing to verify the presence of well-contained interdental bone defects in as many quadrants.

Randomization and Blinding Randomization and blinding included computerized generation of the allocation sequence in random permuted blocks (block randomization) and blinded disbursement of medication. Allocation was performed by assigning the block of sites to study groups according to the specified sequence. Based on the sequence, the first operator selected two sites for each of the following experimental sites; the test site, in which graft (Siloss®) was placed and the control site which was treated by Hydroxyapatite graft only. All the surgeries were performed by a designated operator for the sake of uniformity whereas the relevant readings were recorded by the first operator who was blinded to the nature of the site. The blind was not broken until this clinical trial was completely finished.

Standardization of PPD and CAL PPD and CAL were recorded at the baseline and at the end of 3, 6 and 9 months using a UNC-15 color-coded periodontal probe. An alginate impression was taken and custom acrylic stent limited to the occlusal 2/3rds of the clinical crown were used as fixed reference position (i.e. junction of vertical groove and lower border of the stent). A groove was prepared in the stent to standardize the probing angulation throughout the study period.

Standardization of radiographs Standard digital IOPA radiographs were taken at baseline, 3 and 6 months by the paralleling/long-cone technique at preset parameters using a commercially available RVG (Radiovisiography) system (Kodak RVG 5100® Digital Radiography System, Carestream Health, Rochester, USA). After the imaging plate was placed in the film holder for paralleling technique (XCP Kits for Digital Sensors®, BlueDent, Chennai, India), addition silicon impression material (Elite HD+ Regular Body Normal Set®, Zhermack, Badia Polesine, Italy) was added around the biting surface and allowed to set. This arrangement ensured standardized alignment of the aiming device and the holder ensuring correct positioning of the collimator in subsequent radiographs.

Presurgical protocol Each patient was prepared for surgery with oral hygiene instructions, scaling and root planing at least three months prior to surgery, adjunctive chemical plaque control, and occlusal adjustment was performed, whenever necessary. Patients were re-evaluated to assess clinical parameters and plaque control four weeks after initial therapy.

Study protocol After the interdental areas were probed buccally and lingually/ palatally, the site was considered for study if the average probing pocket depth (PPD) was ≥5 mm. All baseline (on the day of surgery) parameters were recorded before the surgical procedure. The PPD, CAL and site specific plaque scores were recorded at the baseline and at the end of 3, 6 and 9 months. Clinical parameters were recorded using a University of North Carolina no.15 (UNC-15) color-coded Surgical procedure At the start of the surgical procedure, the patients were asked to rinse with 0.2 % chlorhexidine for 1 min. Area subjected to surgery was anesthetized by nerve block/infiltration depending on the surgical site using local anaesthesia. Crevicular incisions were made and the flaps were elevated by means of blunt dissection with the help of a periosteal elevator. The osseous defect was debrided of granulation tissue and the root surface was planed to remove plaque and calculus, until a smooth hard consistency was found. The defect's architecture was confirmed by direct observation and classified based on number of bony walls present. In patients selected for test group, in addition to open flap debridement (OFD), Siloss® bone replacement graft was utilized to fill the defects to the most coronal level of the osseous walls. The required amount of composite alloplast (Siloss®) was dispensed into a sterile dappen dish and mixed with patients own blood and carried to the defect site with an amalgam carrier. The mucoperiosteal flaps were repositioned and secured in place using interrupted sutures. The surgical procedure in control site included open flap debridement followed by placement of hydroxyapatite graft (G-graft®, Saharanpur, UP, India). The surgical area was protected and covered using a periodontal dressing.

Follow-up and postsurgical care Routine postoperative instructions, oral antimicrobials (amoxicillin 500 mg, TID), and analgesics (Diclofenac sodium 50 mg + Paracetamol 325 mg BID) were prescribed for 5 days post operatively and routine post-surgical instructions were explained. Patients were instructed to rinse with 10 ml of 0.2 % chlorhexidine mouthwash twice daily for a week. They were advised to avoid chewing on the surgical site and told not to brush at the site or manipulate it for 10 days one week after the surgery, the dressing and the sutures were removed. Oral hygiene instructions were reinforced. Patients were then monitored at 3, 6, and 9 months. At each of the recall visits, reinforcement of oral hygiene measures, and supragingival scaling if required were performed. At 6 months, all soft tissue measurements were repeated.

Radiographic assessment A single operator evaluated the bone fill by using digital subtraction technique and morphometric area analysis by using specific tools in two image processing software according to a previously described method.

Digital subtraction technique and Morphometric Analysis The radiographs obtained at 3 and 6 months were subtracted from the radiograph taken at the baseline by using commercially available image processing software (Adobe Photoshop® 6.0, Adobe Systems, San Jose, USA). To reduce brightness and contrast variations, both images were adjusted based on the levels and curves in the software. Before digital subtraction, both radiographs were moved in appropriate directions as needed, to reduce geometric distortion. These images were then superimposed and subtracted by selecting the image > calculation> exclusion > new channel tools. The excluded interdental layer was outlined by using the polygonal lasso tool and the layer was copied and saved as a separate joint photographic expert group document at low compression. Morphometric area analysis. After digital subtraction, the digitized and excluded interdental layer was transferred to open source software for area calculation (ImageJ®, Research Services Branch, NIH, Bethesda, Maryland, USA) for area calculation. The layer was converted into a grayscale image, and the measurement scale was set to account for any magnification/reduction of the radiograph because of RVG. The area of the layer was calculated (in mm2) by initially enclosing the entire area with the rectangular selection tool and then by using Analyze > Analyze Particles tool.

Histomorphometric analysis From 3 subjects each from both the groups, bone biopsy specimens were obtained during crown lengthening procedures between 71/2 to 9 months. Briefly, the specimens were immersed in 4% buffered formalin and were subsequently dehydrated in an ascending series of ethyl alcohols. The specimens were then stained using haematoxylin-eosin for light microscopy analysis. 11 and 12 slides were prepared from SILOSS® and HA groups respectively. 10 regions of interest (ROIs) per slide were visualized for mineralized tissue volume by using an Olympus BX 53 microscope at 40X magnification. Before evaluation of bone sections in ImageJ, black and white image masks were created using Adobe Photoshop® according to a technique described by Egan et al.

Calibrating ImageJ To calibrate Image J, a scale bar was placed on one image for each magnification. The file was opened with an image containing a scale bar inserted by the microscope or camera software that acquired the image. The length measured for the scale bar was entered as distance in pixels. The length of the scale bar as labelled by the microscope is entered as known distance and subsequent analysis was measured on this scale.

Quantifying the Mineralized Tissue Volume in ImageJ The bone volume mask file was opened and the total area was selected by Edit> Selection>Select All and Click Analyze>Measure. The "wand tool" and shift key were used to select the black areas. Selecting Analyze>Measure will quantify the mineralized tissue. The Mineralized Tissue Volume was expressed as (mineralized tissue/total area)*100.

Statistical Analysis Site-specific intragroup comparison between various groups was performed using ANOVA followed by multiple comparisons using Bonferroni correction. One-way ANOVA followed by the post hoc test was used for intragroup and intergroup comparison. A p-value of <0.05 was considered statistically significant and p-value of <0.001 was considered as highly significant

ELIGIBILITY:
Inclusion Criteria:

* having at least 2 periodontal pockets ≥5 mm with at least 1 pocket in each quadrant showing radiographic evidence of vertical bone loss were included in the study.

Exclusion Criteria:

* Patients who underwent periodontal therapy in the past 6 months and/or have used antibiotic drugs, antioxidants, and antibacterial mouthwash or medicated toothpastes within 6 months of baseline and smokers were excluded from the study.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth (PPD) and Clinical Attachment Level (CAL) | 9 months
  PPD and CAL were recorded at the baseline and at the end of 3, 6 and 9 months using a UNC-15 color-coded periodontal probe. An alginate impression was taken and custom acrylic stent limited to the occlusal 2/3rds of the clinical crown were used as fixed reference position (i.e. junction of vertical groove and lower border of the stent). A groove was prepared in the stent to standardize the probing angulation throughout the study period.
Digital subtraction technique and Morphometric Analysis | 6 months
  The radiographs obtained at 3 and 6 months were subtracted from the radiograph taken at the baseline by using commercially available image processing software

SECONDARY OUTCOMES:
Quantifying the Mineralized Tissue Volume | 7 to 9 months
  From 3 subjects each from both the groups, bone biopsy specimens were obtained during crown lengthening procedures between 71/2 to 9 months. Briefly, the specimens were immersed in 4% buffered formalin and were subsequently dehydrated in an ascending series of ethyl alcohols. The specimens were then stained using haematoxylin-eosin for light microscopy analysis. 11 and 12 slides were prepared from SILOSS® and HA groups respectively. 10 regions of interest (ROIs) per slide were visualized for mineralized tissue volume by using an Olympus BX 53 microscope at 40X magnification. Before evaluation of bone sections in ImageJ, black and white image masks were created using Adobe Photoshop® according to a technique described by Egan et al.

CONTACTS AND LOCATIONS:
Overall Officials: Rampalli V Chandra, MDS;DNB, Principal Investigator — IEC, SVSIDS, Mahabubnagar
Locations (1):
- SVS Institute of Dental Sciences, Mahabubnagar, Hyderabad, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: No
Data will be shared after publishing the results